CLINICAL TRIAL: NCT01090596
Title: Changes in mRNA Expression Following Exposure to Naproxen
Acronym: Lesions3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Associates of New York, LLP (Other)
Responsible Party: James Aisenberg, MD, Research Associates of New York
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: ResearchANY
Record Dates: First submitted 2010-03-17; First posted 2010-03-22 (Estimated); Last update posted 2010-03-22 (Estimated); Status verified 2010-03

CONDITIONS: Healthy
MeSH Terms: interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naproxen-Treated (Active Comparator)
  Interventions: Drug: Naproxen
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naproxen — 500mg naproxen, twice daily for 7 days
  Arms: Naproxen-Treated
Drug: Placebo — 1 tab,twice a day for a seven days
  Arms: placebo

SUMMARY:
Using tissue samples obtained from a previous study, the effect of naproxen on the gene expression profiles of antral mucosal tissue will be assessed. We hypothesize that there will be distinct changes in the gene expression profiles of samples taken from individuals treated with naproxen versus samples taken from individuals treated with placebo.

DETAILED DESCRIPTION:
We will use microarray technology to quantify the transcriptome-wide changes in gene expression in said-samples.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult between the ages of 18 and 75 inclusive
* Written informed consent prior to undergoing any study procedures
* A physical examination which reveals no clinically significant abnormalities
* Female subjects of childbearing potential must be taking an acceptable form of contraceptive

Exclusion Criteria:

* Any mucosal breaks within 2 cm of pyloric channel seen on baseline endoscopy
* Any GDU or >5 gastroduodenal erosions at baseline endoscopy
* CXB, CPG, ASA, or NS-NSAID use within the prior 2 weeks
* Previous gastrointestinal ulcer
* Hypersensitivity or allergy to NSAIDs, ASA, CPG, CXB or other contraindication to taking treatments
* Baseline complaints of abdominal pain, nausea, and/or cramping
* Any acid blocking medication including antacids, H-2 receptor blocker within the prior 2 weeks, or PPI use within the prior 30 days
* Corticosteroids use within the prior 60 days
* Any documented bleeding tendency
* Has taken warfarin within the prior 60 days
* Three or greater alcoholic beverages daily
* History of cerebro-vascular event

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-04; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Fold Change in Gene Expression | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: James Aisenberg, MD, Principal Investigator — Research Associates of New York